CLINICAL TRIAL: NCT02555449
Title: Disposition of [¹⁴C]-LY3202626 Following Oral Administration in Healthy Male Subjects
Brief Title: A Study of [¹⁴C]-LY3202626 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15566; I7X-EW-LLCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [¹⁴C]-LY3202626 (Experimental): Single oral dose of LY3202626 containing 100 micro curies of radioactivity
  Interventions: Drug: [¹⁴C]-LY3202626

INTERVENTIONS:
Drug: [¹⁴C]-LY3202626 — Administered as solution by mouth

SUMMARY:
The purpose of this study is to measure how much of the specially prepared study drug, LY3202626, containing radiolabeled carbon [¹⁴C] gets into the blood stream and how long it takes the body to get rid of it.

Information about any side effects that may occur will also be collected.

Participants will stay at a clinical research unit (CRU). The study will last about 28 days (check in to follow-up) for each participant.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males, as determined by physical examination, clinical laboratory tests, medical history and electrocardiogram (ECG)
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter squared (kg/m²) inclusive at screening

Exclusion Criteria:

* Have participated in a [¹⁴C]-study within the last 6 months prior to admission for this study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have consumed grapefruits or grapefruit-containing products, Seville oranges or Seville orange-containing products, star fruits or star fruit-containing products within 7 days prior to dosing or intend to consume during the study
* Have a history of constipation or have had acute constipation within 3 weeks prior to admission
* Are currently or have been smokers or users of tobacco or nicotine replacement products within the 3 months prior to admission and/or have positive cotinine at screening or check-in
* Exposure to significant diagnostic, therapeutic, or employment-related radiation within 12 months prior to dosing (e.g., serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- [¹⁴C]-LY3202626: Single 10 milligram (mg) oral dose of LY3202626 containing 100 micro curies of radioactivity
Period: Overall Study
Arm/Group | [¹⁴C]-LY3202626
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- [¹⁴C]-LY3202626: Single oral dose of LY3202626 containing (10 milligrams) 100 micro curies of radioactivity
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 86.40 (6.30)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram/Square Meter (kg/m²)] | 27.90 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Fecal Excretion of Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Fecal excretion of radioactivity over time expressed as a percentage of the total radioactive dose administered.
Time Frame: Predose, 6, 12, 24, 48, 72 Hours At 24 Hour Intervals Until Release Criteria Met
Population: All participants who received the study drug and have evaluable pharmacokinetics (PK) data.
Measure: Mean (Standard Deviation); unit: percentage of the total radioactive dose
Groups:
- [¹⁴C]-LY3202626: Single 10-mg oral dose of LY3202626 containing approximately 100 microcuries of [14C]-LY3202626.
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
percentage of the total radioactive dose | 31.3 (4.24)

2. Primary Outcome: Urinary Excretion of Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Urinary excretion of radioactivity over time was expressed as a percentage of the total radioactive dose administered
Time Frame: Predose, 6, 12, 24, 48, 72 Hours At 24 Hour Intervals Until Release Criteria Met
Population: All participants who received the study drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: percentage of the total radioactive dose
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
percentage of the total radioactive dose | 44.2 (3.70)

3. Secondary Outcome: Plasma Radioactivity Pharmacokinetics Maximum Observed Concentration (Cmax)
Description: Plasma radioactivity pharmacokinetics were measured by the maximum observed concentration (Cmax).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168 Hours At 24 Hour Intervals Until Release Criteria Met
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilter (ng/mL)
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
nanogram/millilter (ng/mL) | 25.2 (16)

4. Secondary Outcome: Plasma Radioactivity Pharmacokinetics Area Under the Concentration-time Curve From Time Zero to Infinity (AUC[0-∞])
Description: Plasma radioactivity pharmacokinetics were measured by the area under the concentration-time curve from time zero to infinity (AUC[0-∞]).
Time Frame: as for outcome 3
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/millilter (ng*h/mL)
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
nanogram*hour/millilter (ng*h/mL) | 1120 (27)

5. Secondary Outcome: Plasma Radioactivity Pharmacokinetics Area Under the Concentration-time Curve From Time Zero to the Last Timepoint With a Measurable Concentration (AUC[0-tlast])
Description: Plasma radioactivity pharmacokinetics were measured by the area under the concentration-time curve from time zero to the last timepoint with a measurable concentration (AUC[0-tlast]).
Time Frame: as for outcome 3
Population: All participants who received the study drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
ng*h/mL | 814 (31)

6. Secondary Outcome: Total Number of Metabolites Representing at Least 10% of the Total Radioactivity in Plasma
Description: Total number of metabolites were identified in at least 10% of the total radioactivity in plasma.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 Hours Postdose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Number; unit: metabolites
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
metabolites | 1

7. Secondary Outcome: Total Number of Metabolites in Excreta (Urine and Feces) That Represent at Least 10% of the Dose of Radioactivity
Description: The total number of metabolites identified in excreta (urine and feces) that represent at least 10% of the dose of radioactivity
Time Frame: From Dosing Until Release Criteria Is Met
Population: All participants who received the study drug and had evaluable PK data.
Measure: Number; unit: metabolites
Arm/Group | [¹⁴C]-LY3202626
Number analyzed (Participants) | 6
metabolites | 2

ADVERSE EVENTS:
Time Frame: From Baseline through End of Study (Up to 2 Months)
Groups:
- [¹⁴C]-LY3202626: Single 10 mg oral dose of LY3202626 containing 100 micro curies of radioactivity
Arm/Group | [¹⁴C]-LY3202626
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [¹⁴C]-LY3202626 (N=6)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days